CLINICAL TRIAL: NCT05119478
Title: Prevalence of Sensitization to Peach and/or Cypress in Potato Sensitized Patients in Occitania
Brief Title: Evaluation of Sensitization to Peach and/or Cypress in Potato Sensitized Patients in a Large Cohort
Acronym: CYPPOT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0612
Record Dates: First submitted 2021-10-27; First posted 2021-11-15 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-10

CONDITIONS: Allergic Rhinitis
Keywords: Cypress; gibberellin-regulated protein; peach; potato; rhinitis
MeSH Terms: conditions — Rhinitis, Allergic; Rhinitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study will be to investigate the prevalence of of sensitization to peach and/or cypress in potato sensitized patients, based on the collection of medical data from patient records consulting in the Allergy Unit of the Arnaud de Villeneuve Hospital.

Some Gibberellin-regulated protein (GRP) in fruits and pollens have been identified as allergen, and peach GRP (peamaclein) has recently emerged as a relevant food allergen in cypress pollen-hypersensitive patients. Multiple fruit allergies might be related to cross-reactivity between GRPs. Peamaclein shares 82% identity with snakin-1 from potato. Thus, because of this hight homology the investigators want to determine the prevalence of cosensitization between these 3 allergens potato, peach and cypress.

ELIGIBILITY:
Inclusion criteria:

* Patients evaluated at the Montpellier University Hospital, Allergy Unit
* children and adult with positive skin prick test to potato from february 2013 to december 2015

Exclusion criteria:

* Patients under legal protection
* Patients under guardianship or under curatorship
* Patients not capable of understanding French

Ages: 2 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients consulting in the Allergy Unit of the Arnaud de Villeneuve Hospital with positive skin prick test to potato
Sampling Method: Non-Probability Sample
Enrollment: 594 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Rate of sensitization to peach and/or cypress in potato-sensitized patients | day 1
  Rate of sensitization to peach and/or cypress in potato-sensitized patients

SECONDARY OUTCOMES:
Rate of of sensitization to peach and/or cypress in potato-sensitized patients | day 1
  Rate of sensitization to peach and/or cypress in potato-sensitized patients (cypress pollen-induced allergic rhinitis or food allergy to peach)

CONTACTS AND LOCATIONS:
Overall Officials: Davide CAIMMI, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC